CLINICAL TRIAL: NCT04172831
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of TNX-102 SL Taken Daily At Bedtime In Patients With Fibromyalgia
Brief Title: A Study To Evaluate The Efficacy And Safety Of TNX-102 SL In Patients With Fibromyalgia
Acronym: RELIEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F304
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Fibromyalgia
Keywords: Pain; Sleep; Fibromyalgia; FM
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablets, 5.6 mg (Experimental): 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 2 weeks then 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablets, 5.6 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
This is a Phase 3, randomized, parallel-group, double-blind, placebo-controlled, 14-week study designed to evaluate the efficacy and safety of TNX-102 SL 5.6 mg (2 x 2.8 mg tablets) taken daily at bedtime for the treatment of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18 to 65 years of age, inclusive.
* The patient has a diagnosis of primary FM as defined by the 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria (American College of Rheumatology Preliminary Diagnostic Criteria)
* The in-clinic 7-day recall NRS average daily pain intensity score at Screening Visit within protocol specified range.

Exclusion Criteria:

* History of or evidence for a diagnosis of borderline personality disorder (BPD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (39):
- United States (39):
  - Tonix Clinical Site, Birmingham, Alabama
  - Tonix Clinical Site, Phoenix, Arizona
  - Tonix Clinical Site, Oceanside, California
  - Tonix Clinical Site, Sacramento, California
  - Tonix Clinical Site, San Diego, California
  - Tonix Clinical Site, Temecula, California
  - Tonix Clinical Site, Cromwell, Connecticut
  - Tonix Clinical Site, Fort Myers, Florida
  - Tonix Clinical Site, Jacksonville, Florida
  - Tonix Clinical Site, North Miami, Florida
  - Tonix Clinical Site, Ocala, Florida
  - Tonix Clinical Site, Orlando, Florida
  - Tonix Clinical Site, Atlanta, Georgia
  - Tonix Clinical Site, Evansville, Indiana
  - Tonix Clinical Site, West Des Moines, Iowa
  - Tonix Clinical Site, Prairie Village, Kansas
  - Tonix Clinical Site, New Orleans, Louisiana
  - Tonix Clinical Site, Boston, Massachusetts
  - Tonix Clinical Site, North Dartmouth, Massachusetts
  - Tonix Clinical Site, Las Vegas, Nevada
  - Tonix Clinical Site, Williamsville, New York
  - Tonix Clinical Site, High Point, North Carolina
  - Tonix Clinical Site, Raleigh, North Carolina
  - Tonix Clinical Site, Fargo, North Dakota
  - Tonix Clinical Site, Cincinnati, Ohio
  - Tonix Clinical Site, Dayton, Ohio
  - Tonix Clinical Site, North Canton, Ohio
  - Tonix Clinical Site, Oklahoma City, Oklahoma
  - Tonix Clinical Site, Tulsa, Oklahoma
  - Tonix Clinical Site, Portland, Oregon
  - Tonix Clinical Site, Allentown, Pennsylvania
  - Tonix Clinical Site, Warwick, Rhode Island
  - Tonix Clinical Site, Chattanooga, Tennessee
  - Tonix Clinical Site, Memphis, Tennessee
  - Tonix Clinical Site, Austin, Texas
  - Tonix Clinical Site, Dallas, Texas
  - Tonix Clinical Site, Salt Lake City, Utah
  - Tonix Clinical Site, Charlottesville, Virginia
  - Tonix Clinical Site, Kenosha, Wisconsin

REFERENCES:
- [Derived] Lederman S, Arnold LM, Vaughn B, Kelley M, Sullivan GM. Efficacy and Safety of Sublingual Cyclobenzaprine for the Treatment of Fibromyalgia: Results From a Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Care Res (Hoboken). 2023 Nov;75(11):2359-2368. doi: 10.1002/acr.25142. Epub 2023 Jul 4. PMID 37165930

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Started | 248 | 255
Completed | 204 | 213
Not Completed | 44 | 42
Not completed — Adverse Event | 21 | 9
Not completed — Lack of Efficacy | 2 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Lost to Follow-up | 4 | 9
Not completed — COVID-19 related crisis | 3 | 3
Not completed — Subject non-compliance | 1 | 1
Not completed — Family emergency | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet | Total
Number analyzed (Participants) | 248 | 255 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.40) | 49.3 (10.16) | 49.6 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 247 | 479
  Male | 16 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 20 | 39
  White | 222 | 216 | 438
  More than one race | 3 | 9 | 12
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 248 | 255 | 503

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 14 in the Numerical Rating Scale (NRS) Weekly Average of Daily Self-reported Average Pain Severity Scores.
Description: Patients provide a daily numeric assessment of their average pain (24-hour recall), via an electronic diary, using an 11-point NRS. Scores range from 0 (no pain) to 10 (worst possible pain).
Time Frame: 14 weeks
Population: Intent to Treat Population (all patient who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -1.9 [-2.1 to -1.7] | -1.5 [-1.7 to -1.3]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.010, Mixed Model Repeated Measures; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.16 — Treatment Difference = TNX-102 - Placebo

2. Secondary Outcome: Number of Patients With a Patient's Global Impression of Change (PGIC) Rating of "Very Much Improved" or "Much Improved"
Description: The PGIC is a fibromyalgia specific validated instrument on a scale of 1 to 7, where a score of 1 indicates the highest level of improvement and a score of 7 indicates a much worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat population (all patient who were randomized). Patients with missing data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
Participants | 93 | 75
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.058, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.99 to 2.10]

3. Secondary Outcome: Change From Baseline to Week 14 in the Fibromyalgia Impact Questionnaire - Revised (FIQR) Symptoms Domain Score
Description: The FIQ-R is a validated questionnaire. Scores on the symptoms domain range from 0 to 100 where a higher score means worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat Population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -18.4 [-20.8 to -16.0] | -14.0 [-16.4 to -11.7]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.007, Mixed Model Repeated Measures; LS Mean Difference = -4.3, 95% CI 2-sided [-7.5 to -1.2], Standard Error of Mean 1.60 — Treatment Difference = TNX-102 - Placebo

4. Secondary Outcome: Change From Baseline to Week 14 in the FIQR Function Domain Score
Description: The FIQ-R is a validated questionnaire. Scores on the function domain range from 0 to 90 where a higher score means worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat Population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -13.6 [-16.1 to -11.2] | -9.3 [-11.7 to -6.8]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.009, Mixed Model Repeated Measures; LS Mean Difference = -4.4, 95% CI 2-sided [-7.7 to -1.1], Standard Error of Mean 1.69 — Treatment Difference = TNX-102 - Placebo

5. Secondary Outcome: Change From Baseline to Week 14 in the Patient Reported Outcomes Measurement Information System (PROMIS) Score for Sleep Disturbance
Description: The PROMIS Sleep disturbance short form 8a consists of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -9.5 [-10.7 to -8.2] | -6.5 [-7.7 to -5.4]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures; LS Mean Difference = -2.9, 95% CI 2-sided [-4.5 to -1.3], Standard Error of Mean 0.82 — Treatment Difference = TNX-102 - Placebo

6. Secondary Outcome: Change From Baseline to Week 14 in the PROMIS Score for Fatigue
Description: The PROMIS fatigue short form 8a consists of 8 questions on a 5 point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -8.0 [-9.1 to -6.9] | -6.2 [-7.4 to -5.0]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.018, Mixed Model Repeated Measures; LS Mean Difference = -1.8, 95% CI 2-sided [-3.3 to -0.3], Standard Error of Mean 0.76 — Treatment Difference = TNX-102 - Placebo

7. Secondary Outcome: Change From Baseline to Week 14 in the Weekly Average of the Daily Diary Assessment of Sleep Quality
Description: Patients provide a daily numeric assessment of their sleep quality for the previous night, via an electronic diary, using an 11-point NRS. Scores range from 0 (best possible sleep) to 10 (worst possible sleep).
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 248 | 255
score on a scale | -2.0 [-2.3 to -1.8] | -1.5 [-1.7 to -1.2]
Statistical Analysis 1: Comparison: TNX-102 SL Tablets, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures; LS Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.17 — Treatment Difference = TNX-102 - Placebo

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | TNX-102 SL Tablets, 5.6 mg | Placebo SL Tablet
All-Cause Mortality (participants affected / at risk) | 0/248 | 0/255
Serious Adverse Events (participants affected / at risk) | 2/248 | 5/255
Other Adverse Events (participants affected / at risk) | 70/248 | 3/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablets, 5.6 mg (N=248) | Placebo SL Tablet (N=255)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Coeliac artery compression syndrome (Gastrointestinal disorders) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypotention (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablets, 5.6 mg (N=248) | Placebo SL Tablet (N=255)
Hypoaesthesia oral (Gastrointestinal disorders) | 43 | 1
Paraesthesia oral (Gastrointestinal disorders) | 14 | 1
Dysguesia (Nervous system disorders) | 13 | 1

LIMITATIONS AND CAVEATS:
Recruitment during COVID-19 pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04172831/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT04172831/SAP_001.pdf